CLINICAL TRIAL: NCT00957151
Title: Evaluation of the Digestive and Metabolic Utilisation of Dietary Protein in Patients With Chronic Pancreatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Avicenne (Other)
Collaborators: Solvay Pharmaceuticals (Industry)
Responsible Party: Pr Benamouzig Robert, AP-HP
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 04007
Record Dates: First submitted 2009-08-11; First posted 2009-08-12 (Estimated); Last update posted 2009-08-12 (Estimated); Status verified 2009-08

CONDITIONS: Chronic Pancreatitis
Keywords: chronic pancreatitis; exocrine pancreatic insufficiency; enzyme therapy; patients with chronic pancreatitis and exocrine pancreatic insufficiency; taking enzyme replacement therapy
MeSH Terms: conditions — Pancreatitis, Chronic; Exocrine Pancreatic Insufficiency | interventions — Pancrelipase

INTERVENTIONS:
Drug: Creon

SUMMARY:
The objective is to evaluate the dietary nitrogen assimilation and metabolic utilisation capability of patients with chronic pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* subjects with chronic pancreatitis and taking enzyme replacement therapy

Exclusion Criteria:

* patients with hepatic impairment
* patients allergic to dairy proteins
* urinary incontinence affecting the measurement of nitrogen metabolism
* digestive disorder affecting the absorption of nutrients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2004-04; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
To measure digestive and metabolic assimilation of dietary proteins in patients with chronic pancreatitis

SECONDARY OUTCOMES:
To determine the efficacy of enzyme therapy

CONTACTS AND LOCATIONS:
Overall Officials: Robert Benamouzig, Pr, Principal Investigator — Department of Gastroenterology